CLINICAL TRIAL: NCT01968889
Title: Diaphragm Function in Patients Acquired Weakness and Neuromyopathy in ICU: Impact on Weaning and Outcome (DIAPH-WEAK ICU)
Brief Title: ICU Acquired Neuromyopathy and Diaphragm Function
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9163
Record Dates: First submitted 2013-08-19; First posted 2013-10-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Critical Illness Myopathy; Respiratory Paralysis
Keywords: Critical illness neuromyopathy; Diaphragm dysfunction; Mechanical ventilation; Weaning; Ultrasound
MeSH Terms: conditions — Respiratory Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Critical illness neuromyopthy: Non invasive phrenic nerve stimulation allowing to measure the twitch airway pressure during airway occlusion
  Interventions: Other: Non invasive phrenic nerve stimulation

INTERVENTIONS:
Other: Non invasive phrenic nerve stimulation — Non invasive phrenic nerve stimulation allowing to measure the twitch airway pressure during airway occlusion

SUMMARY:
Critical illness neuromyopathy is a common disease acquired during ICU stay leading to a deep weakness involving the respiratory muscle work which result in a delayed weaning of mechanical ventilation.

The main objective is to quantify the loss of diaphragm function by measuring the diaphragm force (using the non invasive method by phrenic nerve stimulation allowing to measure the twitch airway pressure during airway occlusion) in a selected population of patients with critical illness neuromyopathy (defined as a MRC score < 48).

The second end points are to evaluate its incidence, the consequences on the patients outcome (extubation success or failure; ICU stay) and to evaluate the relations between diaphragm function (twitch airway pressure during airway occlusion, maximal inspiratory pressure and diaphragm thickness evaluated by ultrasound) and peripheral limbs force (evaluated by the Medical Research Council - MRC score).

DETAILED DESCRIPTION:
Diaphragm function will be assessed through phrenic nerve stimulation allowing to measure the twitch airway pressure during airway occlusion (expressed in cmH2O). It will be assessed during a spontaneous breathing trial for each patient with a known critical illness neuromyopathy. The diaphragm (thickness and course) will be studied by ultrasound assessment as well. Peripheral limbs force will be evaluated by the MRC score. A total of 40 analysable patients will be included.

All these measurements will be made at the time of the spontaneous breathing trial (SBT) during the weaning phase. No modification of the clinical practices of the care should be modified by the study. The twitch airway pressure during airway occlusion will be assessed at the begining of the SBT. The other measurements will be performed 30 mn after the SBT if this one will be well tolerated.

Participants will be followed for the duration of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* MRC score <48
* ready for weaning from mechanical ventilation

Exclusion Criteria:

* previous history of neuromyopathy
* impossibility to perform a magnetic stimulation
* cervical spine injury
* bihemispheric or brain stem lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients acquired weakness and neuromyopathy in ICU
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Twitch tracheal pressure during airway occlusion (expressed in cmH2O) | At the begining of the spontaneous breathing trial
  According the standard of care of weaning process; to evaluate the readiness of the patient to be extubated, the setting of the ventilator should be set at 7 cmH20 PRESSURE SUPPORT VENTILATION (PSV) level and zero end expiratory pressure (PEEP=0) during spontaneous mechanical ventilation to mimic the spontaneous breathing trial (SBT).

SECONDARY OUTCOMES:
extubation success (defined as no need reintubation during the 48h after extubation) | Day 28 after ICU admission
  Participants will be followed until Day 28 after ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Jaber, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Department of Anesthesiology & Critical Care, St Eloi University, Montpellier, France